CLINICAL TRIAL: NCT00554736
Title: A Randomized, Double-blind, Placebo-controlled Trial of Lactobacillus Acidophilus L92 on Markers of Allergic Inflammation by Nasal Provocation With Grass Pollen
Brief Title: Lactobacillus Acidophilus L92 on Markers of Allergic Inflammation by Nasal Provocation With Grass Pollen
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor suspended study do to funding
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200614299-2; 200614299-1 (Other: UC Davis)
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Hayfever
Keywords: Pollen Allergy; Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): In the first phase, subjects with a history of grass pollinosis, with positive skin tests to grass, will be studied out of season and will be randomized to active treatment for 4 months.
  Interventions: Biological: Lactobacillus acidophilus L-92

INTERVENTIONS:
Biological: Lactobacillus acidophilus L-92 — Nasal challenge and acoustic rhinometry will be performed at the first study visit and again at the end of the 4-month supplement period. Standardized perennial ryegrass pollen extract (Lolium perenne) (Hollister-Stier, Inc., Spokane, WA) will be used. Dilutions of the standard product will be made in sterile saline prior to use. The standard product strength is 100,000 BAU/mL. Provocation will start with 100 BAU/mL, delivered as a 100 microliter puff into each nostril nose during breath holding, followed by expiration. Acoustic rhinometry, performed in each nostril, will be recorded at 15 minutes. A change of 30% from baseline in the composite score is considered significant. The dose will be increased every 20 minutes if there is no response. The concentrations used will be 100 BAU, 330 BAU, 1000 BAU, 3300 BAU, 10,000 BAU or 33,000 BAU/mL.

SUMMARY:
This is a placebo controlled double-blind single center study initiated and sponsored by CALPIS, Inc., Japan, and CALPIS U.S.A., Inc., Torrance, CA.

The overall objective of this study is to establish the benefit of a bacterial product, Lactobacillus acidophilus strain L-92 (CALPIS U.S.A., Inc., Torrance, CA), in patients with allergic rhinitis.

DETAILED DESCRIPTION:
The overall objective of this study is to establish the benefit of a bacterial product, Lactobacillus acidophilus strain L-92 (CALPIS U.S.A., Inc., Torrance, CA), in patients with allergic rhinitis. This will be done by noting:

* The threshold dose of pollen extract required on nasal challenge needed to elicit nasal obstruction as measured by acoustic rhinometry pre-treatment, and then comparing the nasal response to the same dose at the end of treatment.
* The dose of pollen extract needed (by progressive dose escalation) to elicit nasal obstruction at the end of treatment if significant nasal obstruction is not reached with the pre-treatment dose.
* Changes in the cytokine and chemokine profile obtained by analysis of the nasal secretion specimens pre- and post-treatment.
* Changes in the cytokine profile of cultured peripheral blood mononuclear cells stimulated with PHA pre- and post-treatment.
* PHADIA ImmunoCAP perennial ryegrass pollen titer pre- and post-treatment.
* The threshold concentration of standardized perennial ryegrass extract to elicit a positive skin prick test pre- and post-treatment
* Total serum IgE pre- and post-

The active product to be used is a tablet made from desiccated Lactobacillus acidophilus strain L-92 and fillers. These bacteria are present in the GI tract of most healthy humans. They are non-pathogenic, and have been used in the food industry for preparation of fermented foods for centuries. They lower the pH of their environment by converting sugar to lactic acid, which inhibits the growth of some pathogens. Lactobacilli are the first genus of bacteria suspected to have health benefits. Most Probiotic studies have been done with live cultures, and indeed there is animal model literature to support greater beneficial immunomodulatory effects of live bacteria over killed organisms. However, some beneficial effects of Lactobacilli are proposed to be due to uptake and processing of cell wall components and bacterial DNA, thus interaction with living bacteria may not be required for all the beneficial effects. However, if a tablet form can deliver live bacteria, in terms of ease of consumption by consumers, it would be preferred by many people, as well as allowing easier blinding of the supplement in clinical trials. The study proposed herein will be the first large study of this product using a live, but desiccated tablet preparation of the bacteria. If this product has a beneficial effect, the fact that it is in a tablet form will greatly benefit consistency in manufacturing, as well as ease storage and ultimate use of the product by consumers.

CALPIS has selected a strain of lactobacilli, L. acidophilus (L92), on the basis of an IgE- lowering effect in experimental studies with mice. This product, in a liquid fermented milk form, has been tested in the following clinical studies:

1. Cedar pollen allergy study (2003). Significant improvement in symptom-medication score was detected (ISHIDA et al BIOSCI. BIOTECH. BIOCHEM. 1652-60, 2005). Product: Liquid fermentation L acidophilus L-92 milk, heat-treated at 75°C for 10 minutes in 100 mL volume.
2. Perennial allergic rhinitis (2002/03). Significant improvement in symptom-medication score was observed (ISHIDA et al J. Dairy Sci. 528-33, 2005). Product: 100 mL heat-treated milk fermented by L acidophilus L-92 (about 3x1010 counts/100 mL)
3. Atopic dermatitis (2005). Improvement in symptom-medication score was detected. Unpublished data. Product: 100 mL fermented milk with L acidophilus L-92.

   An initial study using a desiccated form in tablets has been performed:
4. Artificial pollen allergy study (2005). Improvement in quality of life was noted. Product: desiccated bacteria and fillers in tablets. 20 mg, 60 mg and 180 mg were studied. 180 mg/day was most effective. Unpublished data.

METHODS

PHASE 1

In the first phase, subjects with a history of grass pollinosis, with positive skin tests to grass, will be studied out of season and will be randomized to placebo and active treatment for 4 months. Randomization will be based upon a retrospective Rhinitis Quality of Life Questionnaire regarding their recollection of the worst week of the last pollen season. The intent is to randomize subjects such that the distribution of those with severe versus mild allergy symptoms is equal in both groups. The subjects will be evaluated for their nasal function (patency by acoustic rhinometry) and undergo a nasal provocation test and collection of nasal secretions at the beginning and end of the study. Blood will be drawn and skin tests will be performed at the beginning and end of the study.

Primary Objective:

To assess the efficacy of L-92 versus placebo by comparing the change in nasal obstruction using acoustic rhinometry from the baseline, upon nasal provocation with the same dose of grass pollen extract found to elicit obstruction at enrollment.

Secondary objectives:

1. To compare the change in threshold dose for nasal specific provocation (NPT) test with grass pollen required to elicit nasal obstruction.
2. To compare the change of serum IgE levels to grass pollen (performed by PHADIA ImmunoCAP) and total IgE.
3. To compare the change of cytokines IFN-gamma, IL-2, IL-4, IL-5, IL-9 and IL-13, and the chemokine, eotaxin, in nasal secretion fluid using the same dose of pollen that elicited nasal obstruction at baseline.
4. To compare the change of cytokines IFN-gamma, IL-2, IL-4, IL-5, IL-9 and IL-13 in the supernatant from peripheral blood mononuclear cells (PBMCs) stimulated with PHA pre and post-treatment.

PHASE 2

In the second phase:

Subjects will be given the option to participate for Phase 2 of the study. In this phase, subjects will continue on either placebo or active product throughout the next pollen season, starting in January 2008, and fill out Rhinitis Quality of Life Questionnaires when they pick up the study tablets at the beginning of April, May and June. They will be asked to fill out daily medication/symptom diaries during the first two weeks of May (exact dates subject to change depending on climatic factors). The peak grass pollen season is April through June. Blood will be drawn at a last visit in late June 2008 for specific and total IgE by ImmunoCAP.

ELIGIBILITY:
Inclusion Criteria:

* Each subject qualified by entry criteria history in a brief phone interview will be invited to come to a screening visit. A brief history and targeted physical exam to detect inclusion and exclusion criteria, listed below, will be performed after obtaining informed consent. Then, if the subject still appears eligible, they will undergo allergy skin testing to perennial ryegrass pollen extract as a key inclusion criteria. Skin testing will utilize standard prick techniques with appropriate saline/glycerin controls. The cross sectional measurements of the wheal and flare reaction will be recorded. A positive test will require a wheal >3mm vs the control diluent.

Inclusion Criteria:

* at least a 2-year clinical history of springtime allergic rhinitis
* allergy to grass pollen, defined by positive case history and positive skin prick test
* Males or non-pregnant, non-lactating females who are post-menopausal or naturally or surgically sterile
* Females of childbearing potential should be using acceptable birth control methods
* Patients who are normally active and otherwise judged to be in good health
* Patients must be willing and able to give written informed consent and must provide this consent
* Patients must be willing and able to attend required study visits
* Patients must be able to follow instructions
* Off allergy medication for at least one month prior to study entry (nasal corticosteroids, nasal azelastine, cromolyn sodium, IPRATROPRIUM bromide, antihistamines, leukotriene antagonists)

Exclusion Criteria:

* History of nasal deviation

  * Current cigarette smoker
  * History of allergy symptoms August to January
  * History of nasal polyposis
  * History of asthma
  * Concurrent disease that might complicate or interfere with investigation or evaluation of the study medications
  * Concurrent use of any prohibited medication(s)
  * Chronic or intermittent use of inhaled, oral, intramuscular, intravenous, or potent or super-potent topical corticosteroids
  * Chronic use of long acting antihistamines and other concomitant medications that would affect assessment of the effectiveness of study drug(s)
  * Any systemic disorder that could interfere with the evaluation of the study medication(s)
  * Upper or lower respiratory infection requiring antibiotics within 14 days of the first visit
  * Diagnosis of sinusitis within 30 days of the first Baseline visit
  * Hypersensitivity to the study supplement tablet fillers
  * active or quiescent tuberculosis infection of the respiratory tract
  * nasal septal ulcers, nasal surgery or nasal trauma within 90 days of enrollment
  * Clinical history of anaphylaxis
  * Patients with contraindications for allergy vaccines
  * Clinical history of immunodeficiency, including immunosuppressant therapy
  * Patients with contraindications to adrenaline
  * Subject is taking β-blockers
  * Clinical history of drug or alcohol abuse that would interfere with the patient's participation in the study
  * Clinical history of severe or uncontrolled cardiovascular, hepatic, renal and/or other disease/illness that could be expected to interfere with the study
  * Clinical history, or evidence, of nasolacrimal drainage system malfunction
  * Study site staff who would have access to the clinical study protocol
  * History of immunotherapy with grass pollen extract
  * Participation in any other investigational study within 30 days before entry into this study or concomitantly with this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
The objective is to establish the benefit of Lactobacillus acidophilus strain L-92 in patients with allergic rhinitis. The threshold dose of pollen extract required to elicit nasal obstruction as measured by acoustic rhinometry pre-treatment. | one year

SECONDARY OUTCOMES:
• The dose of pollen extract needed (by progressive dose escalation) to elicit nasal obstruction at the end of treatment if significant nasal obstruction is not reached with the pre-treatment dose. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tong Liu, MD, PhD, Principal Investigator — University of California, Davis

REFERENCES:
- [Background] Ishida Y, Nakamura F, Kanzato H, Sawada D, Hirata H, Nishimura A, Kajimoto O, Fujiwara S. Clinical effects of Lactobacillus acidophilus strain L-92 on perennial allergic rhinitis: a double-blind, placebo-controlled study. J Dairy Sci. 2005 Feb;88(2):527-33. doi: 10.3168/jds.S0022-0302(05)72714-4. PMID 15653517
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical